CLINICAL TRIAL: NCT03957668
Title: Efficacy and Safety of PEG 3350 for Treatment of Chronic Constipation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Collaborators: PT Meiji Indonesia (Unknown)
Responsible Party: Principal Investigator, Murdani Abdullah, Professor, Fakultas Kedokteran Universitas Indonesia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-04-0392
Record Dates: First submitted 2019-05-10; First posted 2019-05-21 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Constipation - Functional
Keywords: PEG 3350; Constipation
MeSH Terms: conditions — Constipation | interventions — polyethylene glycol 3350; Lactulose

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEG 3350 (Experimental): The content of each sachet of PEG 3350 (17 g powder) is dissolved in 240 mL of water, drink it once daily at bedtime, for a duration of 14 days.
  Interventions: Drug: PEG 3350
- Lactulax (Active Comparator): 15 ml of Lactulax syrup (containing 10 g of lactulose) is drunk with 240 ml of water once daily at bedtime, for a duration of 14 days
  Interventions: Drug: Lactulose

INTERVENTIONS:
Drug: PEG 3350 — PEG 3350 17 g once daily for 14 days
  Arms: PEG 3350
Drug: Lactulose — Lactulose 10 g once daily for 14 days
  Arms: Lactulax

SUMMARY:
The aim of this study is to determine the efficacy and safety of PEG 3350 (polyethylene glycol 3350) for short-term treatment of chronic constipation in adults.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged ≥ 18 years.
2. Body Mass Index (BMI) ≥ 18.5
3. Organic bowel disease will be ruled out by Fecal Immunochemical Test (FIT) and/or colonoscopy.
4. Must have ≤ 2 bowel movements during a 7-day qualification period.
5. In otherwise good health as judged by a physical examination and laboratory testing.
6. Not taking medications known to affect bowel function in one week before study.
7. Willing to participate in the study by signing the informed consent.

Exclusion Criteria:

1. Hypersensitive to the study medication.
2. obstructive ileus.
3. Irritable bowel syndrome (IBS) or inflammatory bowel disease (IBD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2019-12-07 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Change of number of bowel movements at 1 week | 7 days
  An increase in the number of bowel movements (defecation) per 7-day period indicates a positive result.
Change of number of bowel movements at 2 weeks | 14 days
  An increase in the number of bowel movements (defecation) per 7-day period indicates a positive result.

SECONDARY OUTCOMES:
Symptom scores at 1 week | 7 days
  * Stool consistency: 0 = hard, 1 = firm, 2 = soft, 3 = loose, 4 = watery (by anamnesis - visual comparison)
  * Stool passage: 0 = strain, 1 = easy, 2 = loss of control (by anamnesis)
  * Cramping and rectal irritation associated with each bowel movement: 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = have to discontinue (by anamnesis)
  * Flatus: 0 = none, 1 = moderate, 2 = occasional, 3 = frequent, 4 = very frequent
Symptom scores at 2 weeks | 14 days
  * Stool consistency: 0 = hard, 1 = firm, 2 = soft, 3 = loose, 4 = watery (by anamnesis - visual comparison)
  * Stool passage: 0 = strain, 1 = easy, 2 = loss of control (by anamnesis)
  * Cramping and rectal irritation associated with each bowel movement: 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = have to discontinue (by anamnesis)
  * Flatus: 0 = none, 1 = moderate, 2 = occasional, 3 = frequent, 4 = very frequent
Overall rating of effectiveness at 1 week | 7 days
  Effective: patients with ≥ 3 bowel movements per 7-day period
Overall rating of effectiveness at 2 weeks | 14 days
  Effective: patients with ≥ 3 bowel movements per 7-day period

OTHER OUTCOMES:
Number of participants with adverse events (AEs) | 7 days, 14 days
  The following adverse events may occur after treatment, thus will be evaluated:
  * Headache
  * Dizziness
  * Fatigue
  * Weakness
  * Nausea
  * Dry mouth
  * Abdominal pain / cramping
  * Flatulence
  * Rectal irritation
  * Diarrhea / watery stool
Number of participants with serious adverse events (SAEs) | 7 days, 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Murdani Abdulah, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (3):
- Indonesia (3):
  - Puskesmas Kelurahan Petamburan, Jakarta, DKI Jakarta
  - RSUPN dr. Cipto Mangunkusumo (Cipto Mangunkusumo Hospital), Jakarta, DKI Jakarta
  - Puskesmas Kelurahan Paseban, Jakarta, DKI Jakarta

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT03957668/Prot_SAP_001.pdf